CLINICAL TRIAL: NCT03595397
Title: Comparative Study of Magnesium Sulfate Versus Fentanyl as Adjuvants to Bupivacaine for Thoracic Epidural Analgesia in Multiple Traumatic Fracture Ribs
Brief Title: Thoracic Epidural Analgesia in Multiple Traumatic Fracture Ribs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed khalid Fathy, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Thoracic Epidural analgesia
Record Dates: First submitted 2018-07-01; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Thoracic Epidural Analgesia, Fracture Ribs
MeSH Terms: interventions — Bupivacaine; Magnesium Sulfate; Fentanyl; Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): 20 patients will receive mid-thoracic epidural analgesia with a loading dose of 8 ml of 0.125% bupivacaine, followed by continuous infusion of 8 ml/hour
  Interventions: Drug: Bupivacaine; Procedure: Thoracic epidural
- Group II (Active Comparator): 20 patients will receive mid-thoracic epidural analgesia with a loading dose of 8 ml mixture of 0.125% bupivacaine and 30 mg/kg magnesium sulfate, followed by continuous infusion of 8 ml/hour of a mixture of 0.125% bupivacaine and 20% magnesium sulfate
  Interventions: Drug: Magnesium Sulfate; Procedure: Thoracic epidural
- Group III (Active Comparator): 20 patients will receive mid-thoracic epidural analgesia with a loading dose of 8 ml of 0.125 bupivacaine and 2 mcg/ml fentanyl, followed by continuous infusion of 8 ml/hour
  Interventions: Drug: Fentanyl; Procedure: Thoracic epidural

INTERVENTIONS:
Drug: Bupivacaine — 20 patients will receive mid-thoracic epidural analgesia with a loading dose of 8 ml of 0.125% bupivacaine, followed by continuous infusion of 8 ml/hour
  Arms: Group I
Drug: Magnesium Sulfate — 20 patients will receive mid-thoracic epidural analgesia with a loading dose of 8 ml mixture of 0.125% bupivacaine and 30 mg/kg Magnesium Sulfate, followed by continuous infusion of 8 ml/hour mixture of 0.125% bupivacaine and 20% Magnesium sulfate
  Other Names: bupivacaine
  Arms: Group II
Drug: Fentanyl — 20 patients will receive mid-thoracic epidural analgesia with a loading dose of 8 ml of 0.125 bupivacaine and 2 mcg/ml fentanyl, followed by continuous infusion of 8 ml/hour.
  Other Names: bupivacaine
  Arms: Group III
Procedure: Thoracic epidural — All patients will receive mid-thoracic epidural analgesia

SUMMARY:
This work aims at comparing the analgesic effect of Thoracic Epidural Magnesium sulfate versus Fentanyl when added as adjuvants to Bupivacaine in patients with multiple traumatic fracture ribs.

DETAILED DESCRIPTION:
Rib fractures are a common condition following trauma with a reported incidence of up to 10% in trauma in general, and up to 39% in blunt chest trauma. Traumatic rib fractures are associated with significant morbidity and mortality, and mortality rates reaching 10-16% has been reported. An estimated one third of patients with traumatic rib fractures develop secondary pulmonary complications with an associated mortality rate as high as 65% . Pain is recognized as a contributing factor to adverse outcome in traumatic rib fractures due to pain-induced inadequate respiratory efforts leading to atelectasis, difficulties in clearing secretions and an increased risk of developing pneumonia. Consequently, adequate analgesia is considered a core intervention in the management of patients with traumatic rib fractures.

There are a variety of ways to manage a patient's pain. Oral analgesic drugs and regional modes are more likely to be used .

Regional analgesia is often supplemented with a small dose of either NSAIDs or opioids and pain reduction is typically strong and immediate. There is little sedation, so evaluation of head and abdominal injuries is easier. A major disadvantage is the technical complexity of the procedures, leading to occasional errors in the administering of the treatments. They can also be painful while the needle is entering (or catheter is being installed), toxicity is a possibility, and the patients require more intensive monitoring and care by the physicians and nurses. There are a variety of modes; the four most common are TEA, thoracic paravertebral block, intercostal block, and intrapleural block. This study focuses on thoracic epidural analgesia.

Narcotic infusions and continuous local anesthetic can be delivered through thoracic or lumbar epidural catheters. Opioid receptors exist in the spinal cord that can alter the perception of pain without needing stimulation of receptors in the brain. After inserting the catheter into this area, local anesthetics and narcotics are administered, blocking the anterior and posterior nerve roots crossing this space. The anesthetic/analgesic agents diffuse across the dura and begin to block sensory nerves. Motor nerves are affected to a lesser degree. It takes a large dose to achieve the desired effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 16 years of age and greater
2. Non-intubated at the time of block placement
3. Traumatic Rib Fractures two or greater
4. Block must be done within 12-24 hours of presentation to the emergency room
5. ASA physical status: I-II

Exclusion Criteria:

1. Patient refusal
2. BMI more than 30 kg/m2
3. Need for mechanical ventilation on admission
4. Hemodynamic instability
5. Haemothorax or Pneumothorax
6. Contraindications of performing blocks as coagulopathy, vertebral column deformities, local infection
7. Traumatic head injury
8. Allergy to local anesthetic agents

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Difference in Pain Scores (Visual Analogue pain scale) | 48 hours
  Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal or vertical scale usually 10 cm or 100 mm length. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale].
  The pain visual analog scale is self completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity.
  After the patient has marked, using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark.
  The scores can be from 0-100.
  A higher score indicates greater pain intensity.
  Based on the distribution of pain, the following cut points on the pain VAS have been recommended:
  No pain (0 -4 mm) Mild pain (5-44 mm) Moderate pain (45-74 mm) Severe pain (75-100 mm)

SECONDARY OUTCOMES:
Development of pulmonary complications: respiratory rate by breath per minute (need for mechanical ventilation) | 48 hours
  By observing respiratory rate of patients using clinical assessment every 1 hour
Assessment of parameters of adequate ventilation and oxygenation: PaO2/FIO2 ratio | 48 hours
  by measuring O2 level in the blood using arterial blood gases every 3 hours
Assessment of parameters of adequate ventilation and oxygenation: PaCO2 in mmHg | 48 hours
  by measuring CO2 level in the blood using arterial blood gases every 3 hours
Changes in heart rate (HR) by beats per minute | 48 hours
  By monitoring patients heart rate every 1 hour
changes in arterial blood pressure (ABP) by mmHg | 48 hours
  By monitoring patients arterial blood pressure using non invasive arterial blood pressure monitoring every 1 hour

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gage A, Rivara F, Wang J, Jurkovich GJ, Arbabi S. The effect of epidural placement in patients after blunt thoracic trauma. J Trauma Acute Care Surg. 2014 Jan;76(1):39-45; discussion 45-6. doi: 10.1097/TA.0b013e3182ab1b08. PMID 24368355
- [Background] Dehghan N, de Mestral C, McKee MD, Schemitsch EH, Nathens A. Flail chest injuries: a review of outcomes and treatment practices from the National Trauma Data Bank. J Trauma Acute Care Surg. 2014 Feb;76(2):462-8. doi: 10.1097/TA.0000000000000086. PMID 24458051
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Wu CL, Jani ND, Perkins FM, Barquist E. Thoracic epidural analgesia versus intravenous patient-controlled analgesia for the treatment of rib fracture pain after motor vehicle crash. J Trauma. 1999 Sep;47(3):564-7. doi: 10.1097/00005373-199909000-00025. PMID 10498316
- [Background] Mackersie RC, Karagianes TG, Hoyt DB, Davis JW. Prospective evaluation of epidural and intravenous administration of fentanyl for pain control and restoration of ventilatory function following multiple rib fractures. J Trauma. 1991 Apr;31(4):443-9; discussion 449-51. PMID 1902264